CLINICAL TRIAL: NCT05675514
Title: Investigation of the Effectiveness of Myofascial Release Technique on Performance Parameters and Injury Risk in Young Basketball: A Randomized Controlled Study
Brief Title: Investigation of the Effectiveness of Myofascial Release Technique in Young Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 09.2022.977
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2022-12

CONDITIONS: Sports Physical Therapy; Myofascial Release Technique; Performance Enhancement; Basketball Players
Keywords: Myofascial Release; Balance; Functional Movement Screen; Performance; Fascia; İnjury Risk
MeSH Terms: interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized with the randomization program called Calculator Soup® (Ashland Global, USA) and divided into 2 groups as intervention and control groups.
  The intervention group; (n=30) at the beginning of the study, after the initial evaluations (demographic information, functional movement screening test (FMS), t agility test, vertical jump test, muscle strength test, muscle viscoelasticity and star balance test) were made, twice a week for 6 weeks, pre-training myofascial release technique will be applied. Final evaluations will be made when the intervention period is over.
  The control group; (n=30) will do their routine training for 6 weeks after the first evaluations (demographic information, FMS, t agility test, vertical jump test, muscle strength test, muscle viscoelasticity and star balance test) and no application will be made. Final evaluations will be made at the end of 6 weeks.
Who Masked: Participant
Masking Description: Participants did not know which group they were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention Group (Experimental): The intervention group; (n=30) at the beginning of the study, after the initial evaluations (demographic information, functional movement screening test (FMS), t agility test, vertical jump test, muscle strength test, muscle viscoelasticity and star balance test) were made, twice a week for 6 weeks, pre-training myofascial release technique will be applied. Final evaluations will be made when the intervention period is over.
  Interventions: Other: Myofascial Release Therapy
- Control Group (No Intervention): The control group; (n=30) will do their routine training for 6 weeks after initial evaluations (demographic information, FMS, t agility test, vertical jump test, muscle strength test, muscle viscoelasticity and star balance test).No action will be taken. Final evaluations will be made at the end of 6 weeks.

INTERVENTIONS:
Other: Myofascial Release Therapy — The increasing number of basketball players also increases the risk of sports-related injuries. Basketball has the highest injury risk of all sports because the game is so powerful and fast moving. Myofascial release therapy; ıt is a form of manual therapy applied on the muscle fascia complex to restore optimal length, reduce pain and improve functions. It is known to be effective in providing rapid relief of pain and tissue sensitivity. By restoring the length and health of the restricted connective tissue with the myofascial release therapy, it aims to relieve pressure on pain sensitive structures such as nerves and blood vessels, as well as improves sports performance.
  Arms: İntervention Group

SUMMARY:
In this study, it is aimed to remove the limitations that cause asymmetry and weak connections in functional movement patterns with myofascial relaxation method to be applied to certain muscles and to remove the obstacles in front of the power factor as a result of its application, to reach the highest efficiency of the athlete's performance and to reduce the risk of injury in the musculoskeletal system.Study; It was planned as a control group (n:30) and an intervention group (n:30). Apart from routine training, the intervention group will be treated twice a week for 6 weeks before the training. On the other hand, no application will be made to the control group other than routine training. The evaluations are; It will be done at the beginning of the study and after the 6-week period.

DETAILED DESCRIPTION:
The study will be randomly divided into two groups and it is planned to include 30 people in each group.

After evaluations (demographic information, functional movement screening test (FMS), t agility test, vertical jump test, muscle strength test, muscle viscoelasticity and star balance test) were made at the beginning of the study in the intervention group (n=30), twice a week for 6 weeks. Myofascial release technique will be performed before the training. Final evaluations will be made 6 weeks after starting the intervention.

The control group (n=30) was excluded from the routine training period for 6 weeks after evaluations (demographic information, functional movement screening test (FMS), T agility test, vertical jump test, muscle strength test, muscle viscoelasticity and star balance test) were made at the beginning of the study. No action will be taken. At the end of 6 weeks, evaluations will be made again.

ELIGIBILITY:
Inclusion Criteria:

* To be playing basketball for at least 6 months
* Being between the ages of 10-16
* Being a man

Exclusion Criteria:

* Having had any surgical operation in the last 6 months.
* Having had a lower/upper extremity injury in the last 3 months.
* A history of anterior cruciate ligament repair
* History of meniscus repair
* History of Achilles tendon repair
* Evaluation intervals to coincide with the pre-season period

Ages: 10 Years to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Functional Movement Screen (FMS) | Change from Baseline FMS score at 6 weeks.
  The Functional Movement Screen (FMS) was designed to identify functional movement deficits and asymmetries that may be predictive of general musculoskeletal conditions and injuries, with an ultimate goal of being able to modify the identified movement deficits through individualized exercise prescription
Vertical Jump Test ( the app My Jump 2) | Change from Baseline jump height score at 6 weeks.
  The MyJump 2 smartphone application is an application that calculates the vertical jump height after determining the time the athlete stays in the air during the jump using the notation method.
Star Excursion Balance Test | Change from Baseline star excursion balance score at 6 weeks.
  Designed to evaluate the dynamic balance in the lower extremity; It is used to monitor progress in rehabilitation, to predict athletes with a high risk of lower extremity injury, and to evaluate deficits that develop after injury.
Muscle Strength Test | Change from Baseline muscle strength test at 6 weeks.
  It is planned to use a digital dynamometer for strength measurements of lower extremity muscles. The dynamometer, whose measurement parameter is set as kilograms of force, is tested with a plastic unit with a force indicator.
  In the evaluations, the subjects are asked to maintain their test positions and to maintain their maximum muscle strength for 3 seconds until they equalize with the opposite force applied by the practitioner.
Agility T Test | Change from Baseline agility t test score at 6 weeks.
  This test is applied to determine the speed of athletes covering distance by changing direction such as forward sprinting, right-left sliding and backward running. The time to finish the test of the athletes is measured with a stopwatch. Each athlete repeats the test twice; The time it takes best will be recorded in seconds.
Muscle Viscoelasticity | Change from Baseline muscle viscoelasticity values at 6 weeks.
  The MyotonPro™ device measures the deformation properties of naturally damped oscillations that occur after mechanical impact on the skin surface (15ms). With this evaluation method; It is possible to measure and evaluate the biomechanical properties of skeletal muscles (muscle tone, stiffness, elasticity) separately from each other in real time with objective, complementary, non-invasive, safe, portable and economical technology.

CONTACTS AND LOCATIONS:
Overall Officials: Gönül Acar, Asst. Prof, Study Director — Marmara University Institute of Health Sciences
Locations (1):
- Vedat GÖKEN, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF), Clinical Study Report (CSR) might be considered to be shared with clinicians studying in the same field one year after the publication of the study.

REFERENCES:
- [Result] Aird L, Samuel D, Stokes M. Quadriceps muscle tone, elasticity and stiffness in older males: reliability and symmetry using the MyotonPRO. Arch Gerontol Geriatr. 2012 Sep-Oct;55(2):e31-9. doi: 10.1016/j.archger.2012.03.005. Epub 2012 Apr 13. PMID 22503549
- [Result] Balsalobre-Fernandez C, Glaister M, Lockey RA. The validity and reliability of an iPhone app for measuring vertical jump performance. J Sports Sci. 2015;33(15):1574-9. doi: 10.1080/02640414.2014.996184. Epub 2015 Jan 2. PMID 25555023
- [Result] Bird SP, Markwick WJ. MUSCULOSKELETAL SCREENING AND FUNCTIONAL TESTING: CONSIDERATIONS FOR BASKETBALL ATHLETES. Int J Sports Phys Ther. 2016 Oct;11(5):784-802. PMID 27757291
- [Result] Cheatham SW, Kolber MJ, Cain M, Lee M. THE EFFECTS OF SELF-MYOFASCIAL RELEASE USING A FOAM ROLL OR ROLLER MASSAGER ON JOINT RANGE OF MOTION, MUSCLE RECOVERY, AND PERFORMANCE: A SYSTEMATIC REVIEW. Int J Sports Phys Ther. 2015 Nov;10(6):827-38. PMID 26618062
- [Result] Cook G, Burton L, Hoogenboom B. Pre-participation screening: the use of fundamental movements as an assessment of function - part 1. N Am J Sports Phys Ther. 2006 May;1(2):62-72. PMID 21522216
- [Result] Cook G, Burton L, Hoogenboom BJ, Voight M. Functional movement screening: the use of fundamental movements as an assessment of function - part 1. Int J Sports Phys Ther. 2014 May;9(3):396-409. PMID 24944860
- [Result] Gribble PA, Hertel J, Plisky P. Using the Star Excursion Balance Test to assess dynamic postural-control deficits and outcomes in lower extremity injury: a literature and systematic review. J Athl Train. 2012 May-Jun;47(3):339-57. doi: 10.4085/1062-6050-47.3.08. PMID 22892416
- [Result] Itotani K, Kawahata K, Takashima W, Mita W, Minematsu H, Fujita H. Myofascial Release of the Hamstrings Improves Physical Performance-A Study of Young Adults. Healthcare (Basel). 2021 Jun 4;9(6):674. doi: 10.3390/healthcare9060674. PMID 34199938
- [Result] Kalichman L, Ben David C. Effect of self-myofascial release on myofascial pain, muscle flexibility, and strength: A narrative review. J Bodyw Mov Ther. 2017 Apr;21(2):446-451. doi: 10.1016/j.jbmt.2016.11.006. Epub 2016 Nov 14. PMID 28532889
- [Result] McKenney K, Elder AS, Elder C, Hutchins A. Myofascial release as a treatment for orthopaedic conditions: a systematic review. J Athl Train. 2013 Jul-Aug;48(4):522-7. doi: 10.4085/1062-6050-48.3.17. Epub 2013 Apr 3. PMID 23725488
- [Result] Monteiro ER, Skarabot J, Vigotsky AD, Brown AF, Gomes TM, Novaes JD. ACUTE EFFECTS OF DIFFERENT SELF-MASSAGE VOLUMES ON THE FMS OVERHEAD DEEP SQUAT PERFORMANCE. Int J Sports Phys Ther. 2017 Feb;12(1):94-104. PMID 28217420
- [Result] Okamoto T, Masuhara M, Ikuta K. Acute effects of self-myofascial release using a foam roller on arterial function. J Strength Cond Res. 2014 Jan;28(1):69-73. doi: 10.1519/JSC.0b013e31829480f5. PMID 23575360
- [Result] Queiroga MR, Lima LS, de Oliveira LEC, Fernandes DZ, Weber VMR, Ferreira SA, Stavinski NGL, Vieira ER. Effect of myofascial release on lower limb range of motion, sit and reach and horizontal jump distance in male university students. J Bodyw Mov Ther. 2021 Jan;25:140-145. doi: 10.1016/j.jbmt.2020.10.013. Epub 2020 Oct 26. PMID 33714485
- [Result] Owoeye OBA, Ghali B, Befus K, Stilling C, Hogg A, Choi J, Palacios-Derflingher L, Pasanen K, Emery CA. Epidemiology of all-complaint injuries in youth basketball. Scand J Med Sci Sports. 2020 Dec;30(12):2466-2476. doi: 10.1111/sms.13813. Epub 2020 Sep 13. PMID 32846028
- [Result] Richman ED, Tyo BM, Nicks CR. Combined Effects of Self-Myofascial Release and Dynamic Stretching on Range of Motion, Jump, Sprint, and Agility Performance. J Strength Cond Res. 2019 Jul;33(7):1795-1803. doi: 10.1519/JSC.0000000000002676. PMID 29912081
- [Result] Schneider S, Peipsi A, Stokes M, Knicker A, Abeln V. Feasibility of monitoring muscle health in microgravity environments using Myoton technology. Med Biol Eng Comput. 2015 Jan;53(1):57-66. doi: 10.1007/s11517-014-1211-5. Epub 2014 Oct 21. PMID 25331739
- [Result] Versteegh T, Beaudet D, Greenbaum M, Hellyer L, Tritton A, Walton D. Evaluating the reliability of a novel neck-strength assessment protocol for healthy adults using self-generated resistance with a hand-held dynamometer. Physiother Can. 2015 Winter;67(1):58-64. doi: 10.3138/ptc.2013-66. PMID 25931654
- [Result] Zhang Q, Trama R, Foure A, Hautier CA. The Immediate Effects of Self-Myofacial Release on Flexibility, Jump Performance and Dynamic Balance Ability. J Hum Kinet. 2020 Oct 31;75:139-148. doi: 10.2478/hukin-2020-0043. eCollection 2020 Oct. PMID 33312302